CLINICAL TRIAL: NCT01941134
Title: Impact of Gastric Bypass Surgery on the Pharmacokinetics of Oral Contraceptive Hormones
Brief Title: Changes in Oral Contraceptive Hormones After Gastric Bypass Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment trouble
Sponsor: Johns Hopkins University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00009641; SFPRF-013-LG (Other: Society for Family Planning)
Record Dates: First submitted 2013-06-12; First posted 2013-09-13 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Bariatric Surgery Candidate; Contraception
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gastric bypass COC (Experimental): This is a before-and-after comparison. Women will enroll prior to planned gastric bypass surgery and complete one cycle of oral contraceptive use and evaluation. There will then be no more study procedures/interventions until 3-4 months after surgery. At that time, women will complete the second cycle of OC use and evaluation. Study participation is then complete.
  Intervention: Ethinyl estradiol-levonorgestrel(EE 20mcg/LNG 150mcg)
  Interventions: Drug: ethinyl estradiol-levonorgestrel

INTERVENTIONS:
Drug: ethinyl estradiol-levonorgestrel — Women will be asked to take a daily ethinyl estradiol-levonorgestrel combined oral contraceptive (COC) for 21 days, beginning 2-3 months pre-operatively, so as to stop at least 30 days before planned surgery date. Then, approximately 3-4 months after surgery, they will again be asked to take a daily pill for 21 days. During these pill cycles, we will collect serum samples and perform ultrasound and cervical mucus assessments on a twice-weekly basis, culminating in an inpatient stay of up to 48 hours in order to obtain more frequent sampling at the end of the pill pack.
  Other Names: EE-LNG oral contraceptive

SUMMARY:
This study will attempt to determine whether having gastric bypass surgery changes the way that the gut absorbs hormones from birth control pills. It is believed that, because gastric bypass surgery causes malabsorption of nutrients and some medications, the levels of birth control hormones after the surgery will be lower than in women before they have the surgery. The investigators will ask several women to take a pack of birth control pills before having bypass surgery, and then another pack several months after surgery. The investigators will measure hormone levels in the blood. The investigators will also measure outcomes that may tell us how well the birth control pills are working, such as ultrasounds of the uterus and ovaries, and examination of the cervix.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo gastric bypass surgery at our institution
* willing to take 2 monthly cycles of the oral contraceptive: one cycle before and one after surgery
* use of Depo-provera within 6 months of enrollment
* Use of implantable or intrauterine contraception
* able to attend multiple study visits

Exclusion Criteria:

* Any contraindication to combined hormonal contraceptive use
* Surgical complications precluding further participation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Serum hormone levels of Ethinyl estradiol and levonorgestrel, as assessed by area under the curve (AUC) | twice weekly x 4 weeks, at 2 separate months: 1 pre-op and one 3-4 months postoperative. Thus, total duration of participation in study will be approximately 7-8 months

SECONDARY OUTCOMES:
Endometrial thickness on transvaginal ultrasound | twice weekly x 4 weeks, at 2 separate months: 1 pre-op and one 3-4 months postoperative. Thus, total duration of participation in study will be approximately 7-8 months
Serum levels of FSH, LH, E and P | twice weekly x 4 weeks, at 2 separate months: 1 pre-op and one 3-4 months postoperative. Thus, total duration of participation in study will be approximately 7-8 months
  Serum levels of Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), estradiol (E) and progesterone (P)
Cervical mucus score | twice weekly x 4 weeks, at 2 separate months: 1 pre-op and one 3-4 months postoperative. Thus, total duration of participation in study will be approximately 7-8 months
  We will assess cervical mucus favorability according to standard criteria.
Presence of ovarian follicles on transvaginal ultrasound | twice weekly x 4 weeks, at 2 separate months: 1 pre-op and one 3-4 months postoperative. Thus, total duration of participation in study will be approximately 7-8 months
  We will assess for and measure ovarian follicles with maximum diameter 10mm or greater

CONTACTS AND LOCATIONS:
Overall Officials: Anne Burke, MD MPH, Principal Investigator — Johns Hopkins University; Kimberly Steele, MD, Principal Investigator — Johns Hopkins University; Roxanne M Jamshidi, MD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States